CLINICAL TRIAL: NCT00183183
Title: Alcohol Screening and Brief Intervention in the Emergency Department
Brief Title: Impact of a Brief Motivational Interview on Drinking Behaviors of At Risk Drinkers Screened in the Emergency Room
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NIAAAASE15123; R21AA015123 (NIH); NIH 5R21AA15123-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Alcohol Abuse
Keywords: Alcohol Abuse; Harm Reduction; Motivational Interviewing; Emergency Department; Risky Drinking; Prevention
MeSH Terms: conditions — Alcoholism; Harm Reduction; Emergencies | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Behavioral: Screening and Brief Intervention

SUMMARY:
Alcohol abuse is associated with injury, chronic illness, absenteeism from work, and social costs to families and communities. The goal of this project is to translate motivational interventions successful in the primary care setting to the Emergency Department (ED) environment by implementing screening, brief intervention and referral to treatment (SBIRT) in order to reduce at-risk drinking among ED patients.

DETAILED DESCRIPTION:
To evaluate the effectiveness of SBIRT in the emergency room setting, ED patients meeting NIAAA criteria for high risk drinking were recruited from 14 sites nationwide (control group-Spring, 2004; intervention group-Summer, 2004). 26% of screened ED patients met inclusion criteria. All enrollees received a list of local referral resources. Intervention group patients also participated in a 15 minute negotiated interview and ED staff referred them directly for treatment if indicated. Enrollees completed 3-month follow-up surveys with a telephone Interactive Voice Response (IVR) system. A total of 1137 patients were enrolled across 14 sites (561 intervention, 576 control), with 62% male, 37% Black, and 38% White, and a mean age of 37. At baseline intervention-i and control-c groups were similar in demographic characteristics and number of drinks on a typical day (mean-i 5.00, mean-c 5.12) and maximum drinks on a given day in the past month (mean-i 7.51, mean-c 7.33). The 3 month follow-up rate was 62% (n=687); the 6 month follow-up rate was 52% (n=567). The 12 month follow up is currently underway.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Communication in English or Spanish
* Met NIAAA criteria for "at-risk drinking":

  * for Men: 15 or more drinks/week, or 5 or more drinks on a single occasion
  * for Women: 8 or more drinks/week, or 4 or more drinks on a single occasion
  * Age 65 or over: 8 or more drinks/week or more than 1 drink per day

Exclusion Criteria:

* Requests detox or already in alcohol treatment program
* Abnormal mental status
* Too ill to give consent
* Unable to provide consent for other reasons
* Suicidal
* Employee or student of site institution (where required)
* Prisoner
* Inability to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1137 (Actual)
Dates: Start 2004-04; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Quantity of drinks per day
Frequency of drinking days per week

SECONDARY OUTCOMES:
Completing alcohol related treatment
Reporting negative alcohol related events

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bernstein, MD, Principal Investigator — Boston University
Locations (15):
- United States (15):
  - Charles R. Drew University of Medicine and Science/Matrin Luther King Hospital, Los Angeles, California
  - University of Southern California Keck School of Medicine / Los Angeles County+University of Southern California Medical Center, Los Angeles, California
  - University of California San Diego Medical Center - Hillcrest, San Diego, California
  - University of Denver/Denver Health Medical Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Section of Emergency Medicine/Yale University School of Medicine, New Haven, Connecticut
  - Howard University/College of Medicine/Department of Pharmacology and Emergency Medicine, Washington D.C., District of Columbia
  - Department of Emergency Medicine Emory University School of Medicine / Emergency Care Center of the Grady Memorial Hospital, Atlanta, Georgia
  - Boston University Medical Center, Boston, Massachusetts
  - Tufts-New England Medical Center Hospital/Tufts University, Boston, Massachusetts
  - University of Michigan Hospital and Health System / Department of Emergency Medicine, Ann Arbor, Michigan
  - Cooper Health/Department of Emergency Medicine at UMNDJ-RWJMS, Camden, New Jersey
  - The University of New Mexico Hospital/Health Sciences Center, Albuquerque, New Mexico
  - Rhode Island Hospital / Brown University / Department of EM and Injury Prevention Center, Providence, Rhode Island
  - University of Virginia Health System, University Hospital, Charlottesville, Virginia